CLINICAL TRIAL: NCT03099876
Title: A Study on Eradication Rate of Triple Therapy Including Low Dose-PPI, Clarithromycin, Amoxicillin According to Treatment Period and CYP2C19 Polymorphisms in H.Pylori Patients
Brief Title: A Study on Eradication Rate of Triple Therapy According to Treatment Period and CYP2C19 Polymorphisms in H.Pylori Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Il-Yang Pharm. Co., Ltd. (Industry)
Responsible Party: Principal Investigator, IL-YANG RA, Il-Yang Pharm. Co., Ltd., Il-Yang Pharm. Co., Ltd.
Other Study IDs: CMC-LDS-ILA02
Record Dates: First submitted 2017-03-28; First posted 2017-04-04 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Helicobacter Pylori Infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Weeks
Biospecimen Retention: Samples With DNA — Blood to anlysis of CYP polymorphism
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 7 days treament group: 7 days of triple therapy (Ilaprazole 10mg, Clarithromycin 500mg Amoxicillin 1000mg B.I.D)
  Interventions: Procedure: treatment period
- 10 days treatment group: 10 days of triple therapy (Ilaprazole 10mg, Clarithromycin 500mg Amoxicillin 1000mg B.I.D)
  Interventions: Procedure: treatment period

INTERVENTIONS:
Procedure: treatment period — 7 days treatment or 10 days treatment

SUMMARY:
This study compared efficacy and safety of basic triple therapy according to treatment period. This study evaluated Effect of CYP2C19 genetic polymorphisms on the efficacy

DETAILED DESCRIPTION:
This study compared efficacy and safety of basic triple therapy including Noltec(Ilaprazole) 10mg, Clapaxine(Clarithromycin) 500mg and Pamoxin Cap(Amoxicillin) 1000mg BID on the first line eradication treatment of H.pylori according to treatment period.

Participants are defined as persons who have endoscopically confirmed on gastric or duodenal ulcer(including scar stage) and gastritis confirmed to be H.pylori positive patients in the UBT test. For 7 days or 10 days Participants treated as basic triple therapy including Noltec(Ilaprazole) 10mg, Clapaxine(Clarithromycin) 500mg and Pamoxin Cap(Amoxicillin) 1000mg BID. After treatment, The healing rate was evaluated in the UBT test at 49±5days from the first day dosing. The investigators would point out the impact of CYP2C19 genotypes on Clarythromycin-based first-line and rescue therapies.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have endoscopically confirmed on gastric, duodenal ulcer(including scar) or gastritis confirmed to be H.pylori positive patients in the biopsy and UBT test.
* Subject who fully understands conditions of clinical trial.
* Subject who agrees to participate and spontaneously sign the ICF

Exclusion Criteria:

* Known hypersensitivity to any component of ilaprazole, Amoxicillin and Levofloxacin
* Subjects who are taking contraindicated medications for experimental and concomitant drug.
* Patients with abnormal levels in the laboratory tests Total Bilirubin, Creatinine> 1.5 times upper limit of normal AST, ALT, Alkaline phosphatase, BUN> 2 times upper limit of normal Administrated of PPI, antibiotic medication within 4 weeks prior to commencement of the study.
* Pregnant and/or lactating women
* Reproductive aged women not using contraception
* Uncontrolled diabetics
* Uncontrolled hypertension
* Uncontrolled liver dysfunction
* Alcoholics
* Subjects with a history of digestive malignancy within 5 years
* Subjects with a history of gastrectomy or esophagectomy Subjects with hereditary diseases such as Galactose intolerance, Lapp lactose deficiency, glucose-galactose malabsorption.
* Subjects participating in a clinical trial before another trial wihin 30 days
* Inconsistence judged subject by researcher

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who visited the hospital
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-12-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
The eradication rate of H.pylori at Day 49±5(or Day 52±5) as assessed by UBT test or Biopsy | Day 49±5(or Day 52±5)
  The eradication rate of H.pylori after 7 days(or 10 days) treatment is defined as those participants who have endoscopically confirmed on gastric or duodenal ulcer(including scar stage) and gastritis confirmed to be H.pylori positive patients in the biopsy or UBT test. The treatment : Noltec(Ilaprazole) 10mg+Pamoxine Cap(Amoxicillin) 1000mg+Clafaxine(Clarithromycin) 500mg was administered twice a day for 7days(or 10days)

SECONDARY OUTCOMES:
The safety of Noltec(Ilaprazole) 10mg BID treatment at Day 49±5(or Day 52±5). Record the number of patients with adverse Events. | Day 49±5(or Day 52±5)
  Record the number of patients with adverse Events. Also Record the symptoms, date, duration, and intensity of Adverse events such.
The eradication rate of H.pylori according to CYP polymorphism of patients. | Day 49±5(or Day 52±5)
  The eradication rate of H.pylori is analyzed accroding to CYP polymorphism: CYP2C19 homo EM, hetero EM, PM
The eradication rate of H.pylori according to stage of disease of patients. | Day 49±5(or Day 52±5)
  The eradication rate of H.pylori is analyzed accroding to stage of disease: active stage, healing stage, scar stage, gastritis.

CONTACTS AND LOCATIONS:
Locations (4):
- South Korea (4):
  - The Catholic Univ. of Korea Daejeon St.Mary Hospital, Daejeon
  - The Chunngnam Univ. General Hospital, Daejeon
  - The Eulji Univ. General Hospital, Daejeon
  - The Konyang Univ. General Hospital, Daejeon